CLINICAL TRIAL: NCT04804761
Title: The Effect of Electroacupuncture (EA) on the Success of Inferior Alveolar Nerve Block (IANB) and Post-operative Pain Relief in Mandibular Molar With Symptomatic Irreversible Pulpitis (SIP) Among Malaysians: A Study Protocol for Randomized Double-Blinded Clinical Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IMU University, Malaysia (Other)
Responsible Party: Principal Investigator, SIN YEN SUAN, Lecturer, IMU University, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCM I/2019(05)
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Symptomatic Irreversible Pulpitis (SIP)
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: Twenty subjects will be recruited from IMU Oral Health Centre, Bukit Jalil who come for endodontic treatment due to symptomatic irreversible pulpitis between April 2020 to April 2022.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The types of treatment, either real or sham EA, will be kept confidential to all parties, including subjects, endodontist, data collector and data analyst, and it will only be reviewed to the acupuncturist right before the EA session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real EA group (Experimental)
  Interventions: Other: Electroacupuncture
- Sham EA group (Sham Comparator)
  Interventions: Other: Electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — Needle insertion on bilateral LI4 HeGu and PC6 NeiGuan and ipsilateral ST6 JiaChe and ST7 XiaGuan (as shown in Table 1), using disposable sterile acupuncture needles (length 25 mm, diameter 0.25 mm; Seirin Corporation, Shizuoka, Japan)

SUMMARY:
Acupuncture is recognized for its pain relief effect. Electroacupuncture(EA) is a form of acupuncture where electric current is passed between pairs of acupuncture needles in order to achieve therapeutic effect. However, there are significantly low number of studies which have discussed the effect of electroacupuncture on dental treatment. Symptomatic irreversible pulpitis is a common condition among dental patients. The success rate of inferior alveolar nerve block before commencing the endodontic treatment of a tooth diagnosed with SIP is reported to be relatively as low as 25%. The aim of this study is to determine the effect of electroacupuncture on the success rate of inferior alveolar nerve block and post-operative pain relief for symptomatic irreversible pulpitis among Malaysians.

DETAILED DESCRIPTION:
A randomized double-blinded clinical pilot study will be conducted in an IMU Oral Health Centre, registered under Malaysia local authority. Convenient stratified blocked random sampling method will be used. Subjects included are those who will undergo endodontic treatment due to SIP between April 2020 to April 2022. 20 subjects are randomly allocated into real and sham acupuncture group. Electroacupuncture on LI4 HeGu, PC6 NeiGuan, ST6 JiaChe and ST7 XiaGuan will be applied on patients for 30 minutes before endodontic treatment. Pain levels are measured with Heft-Parker visual analog scale (HP-VAS) at the time point before and after EA, before and after endodontic treatment, 12 hours, 24 hours and 48 hours after the treatment. For sham acupuncture group, blunted needles which do not penetrate the skin but will only be placed on the skin and stabilised by cotton ball and surgical tape at respective acupuncture points. No manipulation will be conducted for the sham acupuncture group. Patients, endodontist and data analyst are blinded in this study. Data collected will be analysed using Statistical Package for the Social Science (SPSS) version 25.0. Paired T-test will be used to compare the pre-EA and post-EA pain score. T-test will be used to compare the pain scores of real and sham EA groups at each time interval including post-EA, during treatment and post-treatment ; and for induction time of IANBs in real and sham EA groups.

This study will identify the effect of EA on the success rate of IANB and post-operative pain relief for SIP among Malaysian.

ELIGIBILITY:
Inclusion Criteria:

* All Malaysians above the age of 18 years old having a restorable first or second mandibular molar with symptomatic irreversible pulpitis and a history of spontaneous pain presenting with pain level above 54 mm using 170 mm Heft-Parker visual analogue scale (HP-VAS).

Exclusion Criteria:

* Patient with severe systemic disorders, mental disorders, seizures or epilepsy, heart disease, severe clotting disorders, severe periodontal disease or a widening of the periodontal ligament space or periapical radiolucency.
* Patient having a pacemaker.
* Pregnant or lactating women.
* Patient who is true needle phobia [51].
* Patient who has a malignant tumor, wound, infection, lymphedema or fracture at electroacupuncture site.
* Patient who is sensitive to mepivacaine and paracetamol.
* Patient who has a history of treatment with acupuncture, or using any type of medication that could affect the current perception of pain such as tricyclic antidepressants, selective serotonin reuptake inhibitors, analgesics, corticosteroids, or antibiotic at least 24 hours before the endodontic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain levels on HP-VAS after electroacupuncture | Immediately after needle removal
HP-VAS during endodontic procedure | During endodontic procedure

SECONDARY OUTCOMES:
HP-VAS at 12 hours, 24 hours and 48 hours after the treatment | 12 hours, 24 hours and 48 hours after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yen Suan Sin, Principal Investigator — IMU University, Malaysia
Locations (1):
- International Medical University, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] European Society of Endodontology. Quality guidelines for endodontic treatment: consensus report of the European Society of Endodontology. Int Endod J. 2006 Dec;39(12):921-30. doi: 10.1111/j.1365-2591.2006.01180.x. PMID 17180780
- [Background] Erdem Hepsenoglu Y, Eyuboglu TF, Ozcan M. Postoperative Pain Intensity after Single- versus Two-visit Nonsurgical Endodontic Retreatment: A Randomized Clinical Trial. J Endod. 2018 Sep;44(9):1339-1346. doi: 10.1016/j.joen.2018.05.017. Epub 2018 Jul 24. PMID 30054099
- [Background] Aggarwal V, Singla M, Miglani S, Kohli S. Comparative Evaluation of Mental Incisal Nerve Block, Inferior Alveolar Nerve Block, and Their Combination on the Anesthetic Success Rate in Symptomatic Mandibular Premolars: A Randomized Double-blind Clinical Trial. J Endod. 2016 Jun;42(6):843-5. doi: 10.1016/j.joen.2016.02.015. Epub 2016 Apr 14. PMID 27086046
- [Background] Click V, Drum M, Reader A, Nusstein J, Beck M. Evaluation of the Gow-Gates and Vazirani-Akinosi techniques in patients with symptomatic irreversible pulpitis: a prospective randomized study. J Endod. 2015 Jan;41(1):16-21. doi: 10.1016/j.joen.2014.09.010. Epub 2014 Nov 6. PMID 25442724
- [Background] Drum M, Reader A, Nusstein J, Fowler S. Successful pulpal anesthesia for symptomatic irreversible pulpitis. J Am Dent Assoc. 2017 Apr;148(4):267-271. doi: 10.1016/j.adaj.2017.01.002. Epub 2017 Feb 9. PMID 28190451
- [Background] Fowler S, Drum M, Reader A, Beck M. Anesthetic Success of an Inferior Alveolar Nerve Block and Supplemental Articaine Buccal Infiltration for Molars and Premolars in Patients with Symptomatic Irreversible Pulpitis. J Endod. 2016 Mar;42(3):390-2. doi: 10.1016/j.joen.2015.12.025. Epub 2016 Jan 28. PMID 26831048
- [Background] Kung J, McDonagh M, Sedgley CM. Does Articaine Provide an Advantage over Lidocaine in Patients with Symptomatic Irreversible Pulpitis? A Systematic Review and Meta-analysis. J Endod. 2015 Nov;41(11):1784-94. doi: 10.1016/j.joen.2015.07.001. Epub 2015 Aug 17. PMID 26293174
- [Background] Topcuoglu HS, Arslan H, Topcuoglu G, Demirbuga S. The Effect of Cryotherapy Application on the Success Rate of Inferior Alveolar Nerve Block in Patients with Symptomatic Irreversible Pulpitis. J Endod. 2019 Aug;45(8):965-969. doi: 10.1016/j.joen.2019.05.001. Epub 2019 Jun 14. PMID 31204040
- [Background] Saatchi M, Khademi A, Baghaei B, Noormohammadi H. Effect of sodium bicarbonate-buffered lidocaine on the success of inferior alveolar nerve block for teeth with symptomatic irreversible pulpitis: a prospective, randomized double-blind study. J Endod. 2015 Jan;41(1):33-5. doi: 10.1016/j.joen.2014.09.011. Epub 2014 Oct 31. PMID 25442722
- [Background] Dianat O, Mozayeni MA, Layeghnejad MK, Shojaeian S. The efficacy of supplemental intraseptal and buccal infiltration anesthesia in mandibular molars of patients with symptomatic irreversible pulpitis. Clin Oral Investig. 2020 Mar;24(3):1281-1286. doi: 10.1007/s00784-019-03006-8. Epub 2019 Jul 13. PMID 31302768
- [Background] Nagendrababu V, Pulikkotil SJ, Jinatongthai P, Veettil SK, Teerawattanapong N, Gutmann JL. Efficacy and Safety of Oral Premedication on Pain after Nonsurgical Root Canal Treatment: A Systematic Review and Network Meta-analysis of Randomized Controlled Trials. J Endod. 2019 Apr;45(4):364-371. doi: 10.1016/j.joen.2018.10.016. Epub 2019 Feb 6. PMID 30737050
- [Background] Aminoshariae A, Kulild JC, Donaldson M. Short-term use of nonsteroidal anti-inflammatory drugs and adverse effects: An updated systematic review. J Am Dent Assoc. 2016 Feb;147(2):98-110. doi: 10.1016/j.adaj.2015.07.020. Epub 2015 Nov 6. PMID 26562732
- [Background] Sostres C, Gargallo CJ, Arroyo MT, Lanas A. Adverse effects of non-steroidal anti-inflammatory drugs (NSAIDs, aspirin and coxibs) on upper gastrointestinal tract. Best Pract Res Clin Gastroenterol. 2010 Apr;24(2):121-32. doi: 10.1016/j.bpg.2009.11.005. PMID 20227026
- [Background] Mandegaran R, Conway C, Elton C. Lower gastrointestinal adverse effects of NSAIDS: an extreme example of a common problem. BMJ Case Rep. 2013 Feb 20;2013:bcr2012008274. doi: 10.1136/bcr-2012-008274. PMID 23429022
- [Background] Carrotte P. Endodontics: Part 3. Treatment of endodontic emergencies. Br Dent J. 2004 Sep 25;197(6):299-305. doi: 10.1038/sj.bdj.4811641. PMID 15454989
- [Background] Pak JG, White SN. Pain prevalence and severity before, during, and after root canal treatment: a systematic review. J Endod. 2011 Apr;37(4):429-38. doi: 10.1016/j.joen.2010.12.016. PMID 21419285
- [Background] Arias A, de la Macorra JC, Hidalgo JJ, Azabal M. Predictive models of pain following root canal treatment: a prospective clinical study. Int Endod J. 2013 Aug;46(8):784-93. doi: 10.1111/iej.12059. Epub 2013 Feb 12. PMID 23402273
- [Background] Simpson M, Drum M, Nusstein J, Reader A, Beck M. Effect of combination of preoperative ibuprofen/acetaminophen on the success of the inferior alveolar nerve block in patients with symptomatic irreversible pulpitis. J Endod. 2011 May;37(5):593-7. doi: 10.1016/j.joen.2011.02.015. Epub 2011 Mar 22. PMID 21496654
- [Background] Parirokh M, Ashouri R, Rekabi AR, Nakhaee N, Pardakhti A, Askarifard S, Abbott PV. The effect of premedication with ibuprofen and indomethacin on the success of inferior alveolar nerve block for teeth with irreversible pulpitis. J Endod. 2010 Sep;36(9):1450-4. doi: 10.1016/j.joen.2010.05.007. Epub 2010 Jul 3. PMID 20728707
- [Background] Bushra R, Aslam N. An overview of clinical pharmacology of Ibuprofen. Oman Med J. 2010 Jul;25(3):155-1661. doi: 10.5001/omj.2010.49. PMID 22043330
- [Background] Hargreaves K, Abbott PV. Drugs for pain management in dentistry. Aust Dent J. 2005 Dec;50(4 Suppl 2):S14-22. doi: 10.1111/j.1834-7819.2005.tb00378.x. PMID 16416713
- [Background] Jalali S, Moradi Majd N, Torabi S, Habibi M, Homayouni H, Mohammadi N. The Effect of Acupuncture on the Success of Inferior Alveolar Nerve Block for Teeth with Symptomatic Irreversible Pulpitis: A Triple-blind Randomized Clinical Trial. J Endod. 2015 Sep;41(9):1397-402. doi: 10.1016/j.joen.2015.04.026. Epub 2015 Jun 16. PMID 26092771
- See also: Related Info — https://www.aae.org/specialty/clinical-resources/glossary-endodontic-terms/
- See also: Related Info — https://www.elsevier.com/books/ten-cates-oral-histology/nanci/978-0-323-48524-1
- See also: Related Info — https://www.aae.org/patients/root-canal-treatment/what-is-a-root-canal/root-canal-explained/
- See also: Related Info — https://www.researchgate.net/publication/316875589_Prevalence_of_endodontic_diseases_An_epidemiological_evaluation_in_a_Brazilian_subpopulation
- See also: Related Info — https://www.researchgate.net/publication/51589734_Diagnostic_and_clinical_factors_associated_with_pulpal_and_periapical_pain
- See also: Related Info — https://www.researchgate.net/publication/257736619_Comparison_of_the_oral_health-related_quality_of_life_and_dental_pain_in_symptomatic_irreversible_pulpitis_and_pericoronitis
- See also: Related Info — https://www.who.int/traditional-complementary-integrative-medicine/en/
- See also: Related Info — http://www.pharmnet.com.cn/tcm/zjdq/jzzj/100047.html
- See also: Related Info — https://www.amazon.com/Science-Acupuncture-Moxibustion-Jianqiao-Fang/dp/7513218773
- See also: Related Info — https://www.cnki.net/kcms/doi/10.13703/j.0255-2930.2017.06.019.html
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2396469/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6416101/
- See also: Related Info — http://www.electroacupunctureknowledge.com/
- See also: Related Info — https://www.ccaom.org/images/ccaom/Documents/7th_Edition_Manual_Chinese_June_2017.pdf
- See also: Related Info — http://kns.cnki.net/kcms/detail/detail.aspx?filename=GYYX200201007&dbcode=CJFQ&dbname=cjfd2002&v